CLINICAL TRIAL: NCT04542031
Title: COVID-19 Prevalence in a Single Large UK Rheumatology Centre and the Impact on Quality of Life From Stringent Social Distancing
Brief Title: COVID-19 in a Single Large UK Rheumatology Centre and Impact on QOL
Acronym: CRISP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Royal Wolverhampton Hospitals NHS Trust (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2020COV113
Record Dates: First submitted 2020-09-07; First posted 2020-09-09 (Actual); Last update posted 2025-01-06 (Actual); Status verified 2025-01

CONDITIONS: Covid19; Rheumatic Diseases
MeSH Terms: conditions — COVID-19; Rheumatic Diseases | interventions — Surveys and Questionnaires

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Survey (Other): Survey to be distributed at 6 and 12 months
  Interventions: Other: Questionnaire

INTERVENTIONS:
Other: Questionnaire — Questionnaire to be completed at 6 and 12 months

SUMMARY:
The COVID-19 pandemic represents a threat to rheumatology patients. National advice for patients to 'shield' is based on risk stratification of therapies and other risk factors. While the epidemiology of COVID-19 in the rheumatological population is largely unknown large case registries are beginning to show potential drug treatment interactions. Strict self-isolation (shielding) has been recommended for those deemed 'high risk' although its impact on the likelihood of COVID-19 infection and health related quality of life (HRQoL) is unclear.

The study aims to explore how this unprecedented situation has impacted the Trust patients primarily evaluating prevalence of the infection, effect of stringent social distancing (shielding) and Quality of Life (QOL). This will be done via a voluntary questionnaire, sent via text messaging at 6 and 12 months.

ELIGIBILITY:
Inclusion Criteria:

* All rheumatology patients under active follow up at the Royal Wolverhampton Trust with a validated mobile telephone number

Exclusion Criteria:

* Patients without a validated mobile phone number linked to their hospital record

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1010 (Actual)
Dates: Start 2020-12-14 (Actual); Primary Completion 2022-02-01 (Actual); Study Completion 2022-02-01 (Actual)

PRIMARY OUTCOMES:
Prevalence of COVID 19 | 1 year
  percentage of cases
Mortality rates from COVID 19 | 1 year
  number of deaths per 1000 individuals
Health related quality of life - Short Form 12 | 1 year
  mental and physical component scores through patient reported outcomes. Normative score set at 50 with minimum score being 0 and maximum score being 100. Scores >50 indicate better mental or physical health than the mean. Scores <50 indicate worse mental or physical health than the mean

CONTACTS AND LOCATIONS:
Overall Officials: James Bateman, Principal Investigator — The Royal Wolverhampton NHS Trust
Locations (1):
- The Royal Wolverhampton NHS Trust, Wolverhampton, West Midlands, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Cox N, Raizada SR, Barkham N, Venkatachalam S, Sheeran TP, Adizie T, Sapkota H, Scott IC, Muller S, Bateman J. The impact of the COVID-19 pandemic and stringent social distancing measures on health-related quality of life and COVID-19 infection rates in patients with rheumatic disease: a longitudinal analysis through the pandemic. Rheumatol Adv Pract. 2023 Jan 16;7(1):rkad009. doi: 10.1093/rap/rkad009. eCollection 2023. PMID 36751643